CLINICAL TRIAL: NCT02044731
Title: Impact of a Childhood Obesity Intervention for African American Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-07-4508 B; 033728B (Other Grant/Funding Number: Safeway Foundation)
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Obesity; Overweight
Keywords: Schools; Pediatrics; Obesity; Overweight; Intervention Studies; African Americans; Family; Body mass index
MeSH Terms: conditions — Obesity; Overweight | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Family group sessions (Experimental): Active and Healthy Families
  Interventions: Behavioral: Active and Healthy Families

INTERVENTIONS:
Behavioral: Active and Healthy Families — A pediatric overweight/obesity intervention delivered through five bi-weekly family-based group sessions.

SUMMARY:
The purpose of this study is to evaluate the impact on body mass index (BMI) of a 5-session childhood obesity intervention for African American families among children aged 5-12 years. We hypothesize that children participating in the program will experience a reduction in BMI.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than or equal to the 85th percentile for age and sex
* Attends an elementary school in the Pittsburg Unified School District in California
* Parent of child meeting above criteria

Exclusion Criteria:

-

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Body mass index (BMI) | Baseline and at week 10
  Change in BMI will be calculated from measured height and weight

SECONDARY OUTCOMES:
Blood pressure | Baseline and at week 10
  Change will be calculated based on measured blood pressure

OTHER OUTCOMES:
Parent weight | Baseline and at week 10
  Change will be calculated based on measured weight of parent
Parent reported behaviors | Baseline and at 10 weeks
  Survey responses on parenting and child's dietary, physical activity, and screen time behaviors.
Parent blood pressure | Baseline and at week 10

CONTACTS AND LOCATIONS:
Overall Officials: Kristine A Madsen, MD, Principal Investigator — University of California, Berkeley
Locations (1):
- Parkside Elementary School, Pittsburg, California, United States